CLINICAL TRIAL: NCT05865275
Title: The Use of Diode Low-power Laser Therapy Before of In-office Bleaching to Prevent the Bleaching-induced Tooth Sensitivity. A Clinical Study
Brief Title: Diode Low-power Laser Before In-office Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, felice femiano, associate Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2023-04-29; First posted 2023-05-18 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Tooth Sensitivity
Keywords: in-office bleaching; tooth sensitivity; low-level laser; therapy (LLLT); pain.
MeSH Terms: conditions — Dentin Sensitivity; Pain

STUDY DESIGN:
Intervention Model Description: A randomized double-blind and placebo-controlled clinical trial study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * an investigator was employed for patient recruitment and to perform preliminary sensitivity tests at baseline for all selected patients (baseline)
  * a non-clinical investigator was used to divide the patients into two study groups using random distribution software.
  The laser procedure and the whitening procedure were performed by two different clinical operators who were not aware of the organization of the two study groups.
  Subsequently, the first operator, already employed to collect scores in baseline, and who was unaware of the assigned clinical protocols, underwent again all participants of the study to sensitivity Test asking them to record the degree of dental sensitivity, for each bleached tooth, perceived from immediately, to 1 h, to 24 h, and 48 h after the end of bleaching treatment using the score.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): it is the group for testing the effectiveness of low power of a diode laser on the onset of dental sensitivity
  Interventions: Device: Low-level laser treatment; Other: tooth bleaching procedure
- Placebo group (Placebo Comparator): this represents the control group with tooth bleaching without preliminary laser treatment
  Interventions: Other: tooth bleaching procedure

INTERVENTIONS:
Device: Low-level laser treatment — a single preliminary treatment for a few seconds for each tooth using low level diode laser before of tooth bleaching could reduce risk to arise of tooth sensitivity
  Other Names: use of low-power diode laser before tooth bleaching
  Arms: Test group
Other: tooth bleaching procedure — The gingival tissues of the teeth to be bleached were isolated from the bleaching gel using a light-cured resin dam (OpalDam Kit, Ultradent; Milan, Italy). A 38 % ready-to-use Hydrogen peroxide-containing gel (The Smile® Strong, Italy) was applied from the first premolar right to the first premolar left of both jaws for a total period of 20 minutes for a 1 single whitening session.

SUMMARY:
Background: The aim of study was to investigate the effectiveness of low-level laser therapy (LLLT) use before in-office bleaching to prevent risk and intensity of tooth sensitivity.

Methods: thirty patients were selected for this clinical trial. Before bleaching procedures with 38 % hydrogen peroxide, the participants were randomly divided into two groups of 15 subjects. Test group: the patients teeth received a preliminary LLLT procedure by an 810 nm diode laser with 0.5 Watt for 30 s for an energy density of 15 J/cm2 and a group placebo: the patients received the same preliminary LLLT but with the device switch off. All patients were instructed to report their cold sensitivity experiences immediately, 1 h, 24 h, and 48 h after the end of bleaching by a visual analog scale score between 0-10.

DETAILED DESCRIPTION:
Materials and methods The sample used for this study was of 30 subjects with explicit request for teeth whitening and was conducted in agreement with a randomized double-blind and placebo controlled clinical trial. This search was led in accordance with the ethical standards of the committee responsible for human experimentation (institutional and national), and with the Helsinki Declaration of 1975, as revised in 2013. Only patients at least 18 years old with teeth of a shade darker than C2, using the shade guide of Vita Classical A1-D4®- Germany, were recruited. All patients were in good general health with maxillary and mandibular anterior teeth without caries, visible defects, and any restoration. Subjects who exhibited a negative vitality test for any teeth, from 1.4 to 2.4, were excluded from the study. Patients who used analgesics, anti-inflammatory, or antioxidant medicine to therapeutic purposes and those with smoking habits, also were excluded from the study as well as patients with bruxism habits or with any pathologic defect such as gingival recession or dentin exposure. None of the patients recruited reported symptoms attributable to dental sensitivity. Two weeks before the bleaching treatment, the participants underwent professional oral hygiene and received oral hygiene instructions to brush their teeth twice per day with a similar toothbrush and toothpaste during the research time. Each patient was informed, verbally and in writing, about the treatment procedures and was asked to sign an informed consent document before the study commencement. All the teeth from 1.4 to 2.4 of each patient that had to be subjected to whitening treatment were evaluated for dental sensitivity by means of the cool sensitivity test (baseline).

Cold sensitivity Test (CST): The degree of tooth sensitivity was determined using an air stimulus deﬁned as a 3 s cold air blast (temperature range of 19-20° C) at a distance of 2-3 mm from the test site. Each tooth under examination was isolated using cotton rolls and by shielding the neighboring teeth with the gloved ﬁngers of the operator. All patients were asked to report their degree of sensitivity for each tooth after the CST employing a visual analog scale (VAS) to objectify the degree of intensity of pain/discomfort felt, consisting of a 100-mm horizontal line on a sheet of paper with 0-10 points where the ends were represented from 0 (the left side) indicating no pain/discomfort and 10 (the right side) representing the worst possible pain never warned [14].

Patients reporting VAS values greater than 4 for at least one tooth were excluded from the study.

The in-office bleaching procedure The thirty patients selected have randomly divided into two groups (n=15) using a Random Number Generator Software by a not-clinician investigator. The mean age of the patients was similar in the two study groups (test group 23.4 ± 5.8 and placebo group 5.5 ± 6.2), as well as there was no significant difference in the sex of the participants between the two groups (8 and 7 females respectively in test and placebo group).

* Test group: all teeth to be whitened of each patient, before bleaching, received an irradiation procedure by a LLLT using a diode laser (Soft Touch; 810 nm, 5 W, Creation). The laser probe (a fiber of 400 µm diameter) was positioned in contact mode with the enamel of the tooth to be irradiated for 30 s in continuous-wave using 0.5 W, with horizontal and vertical moving to cover the whole area. Each tooth received an energy density of 15 J/cm2. Subsequently each patient underwent the teeth whitening procedure using the protocol recommended by the product manufacturer. The gingival tissues of the teeth to be bleached were isolated from the bleaching gel using a light-cured resin dam (OpalDam Kit, Ultradent; Corsico- MILAN, Italy). A 38 % ready-to-use Hydrogen peroxide-containing gel (The Smile® Strong, Italy) was applied from the first premolar right to the first premolar left of both jaws for a total period of 20 minutes for a 1 single whitening session.
* Placebo group: all teeth to be whitened of each patient, before bleaching, to avoid interference psychological of patients on outcomes of study, received a preventive laser procedure applying the identical parameters used for group test except the device was kept in idle mode. Subsequently he teeth whitening procedure was identical to that of the test group.

Following the bleaching treatment, the gel was rinsed off. The laser procedure and the whitening procedure were performed by two different clinical operators who were not aware of the organization of the two study groups.

Subsequently, the first operator, already employed to collect VAS score in baseline, and who was unaware of the assigned clinical protocols, underwent again all participants of the study to CST asking them to record the degree of dental sensitivity, for each bleached tooth, perceived from immediately, to 1 h, to 24 h, and to 48 h after the end of bleaching treatment using the VAS score.

Statistical analysis To quantify the cold discomfort experience for each patient a single VAS value was considered, obtained from the sum of the individual VAS values from each tooth exposed to cold test. While, for the comparsion of discomfort between the two groups, the total VAS score of each group was used, resulting from the sum of the VAS values of each patient collected at the different study times. The VAS values of each group was confronted with each other and also compared with the baseline value of reference at different study times.The statistical analysis was performed with GraphPad Prism software version 9 (by Dotmatics, San Diego CALIFORNIA, USA.) The significance level for all tests was predetermined at p< 0.05.

Results All 30 participants completed the study. The table 1 shows the total value VAS (mean and standard deviation, SD) for each study group at different time points of the clinical trial. The comparison of the total VAS scores for each group study within the same study time revealed statistically significant values using the Wilcoxon signed-rank test in times of immediately, after 1h, and after 24 h while there was no significant difference for the VAS values 48 h after whitening treatment (Table 1 and figure 1). The comparison of VAS score of each group with the corresponding value at baseline time shows high significance for both groups in immediately and only with the equivalent VAS value of placebo group after 1 h and 24 h after whitening.

ELIGIBILITY:
Inclusion Criteria:

* patients with teeth of a shade darker than C2, using the shade guide of Vita Classical A1-D4®- Germany
* patients in good general health with maxillary and mandibular anterior teeth without caries, visible defects, and any restoration.

Exclusion Criteria:

* Subjects who exhibited a negative vitality test for any teeth, from 1.4 to 2.4,
* Patients who used analgesics, anti-inflammatory, or antioxidant medicine for therapeutic purposes and those with smoking habits, also were excluded from the study as well as patients with bruxism habits or with any pathologic defect such as gingival recession or dentin exposure.
* Patients with symptoms attributable to dental sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
baseline | time 0
  The total scores in each study group of dental hypersensitivity
Immediately | Immediately after the end of bleaching treatment
  The total scores in each study group of dental hypersensitivity
After 1 hour | to 1 h after the end of bleaching treatment
  The total scores in each study group of dental hypersensitivity
After 24 hours | to 24 h after the end of bleaching treatment
  The total scores in each study group of dental hypersensitivity
After 48 hours | to 48 h after the end of bleaching treatment
  The total scores in each study group of dental hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: rossella femiano, Principal Investigator — University of Campania Luigi Vanvitelli; vincenzo grassia, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- Multidisciplinary Department of Medical-Surgical and Dental Specialties, University of study of Campania, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD will be registered in an exel file and the same will be upload on an virtual drive as dropbox or google drive
Supporting Information: Study Protocol
Time Frame: The data will be avaible after article publication with no time limitation
Access Criteria: all data will be avaible contacting corresponding author indicated in the published article

REFERENCES:
- [Background] Ahrari F, Akbari M, Mohammadpour S, Forghani M. The efficacy of laser-assisted in-office bleaching and home bleaching on sound and demineralized enamel. Laser Ther. 2015 Dec 30;24(4):257-64. doi: 10.5978/islsm.15-OR-15. PMID 26877590
- [Background] Naghsh N, Kachuie M, Bijari M, Birang R. Evaluation of the effects of 980 and 810-nm high-level diode lasers in treating dentin hypersensitivity: A double-blinded randomized clinical trial. Dent Res J (Isfahan). 2022 Nov 17;19:96. eCollection 2022. PMID 36605144
- [Background] Mendez Romero JM, Villasanti Torales UA, Villalba Martinez CJ. Efficacy of laser application in dental bleaching: A randomized clinical controlled trial. Am J Dent. 2020 Apr;33(2):79-82. PMID 32259412